CLINICAL TRIAL: NCT03518944
Title: Establishing of an Early Warming System of Premature Ovarian Insufficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2017-197
Record Dates: First submitted 2018-03-28; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2017-08

CONDITIONS: Primary Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- occult premature ovarian insufficiency: Serum FSH levels ≥10mIU/ml/ serum AMH levels ≤1.0pg/ml/ AFC ≤5, on at least two occasion >4 weeks apart

SUMMARY:
Premature ovarian insufficiency (POI) is a clinical syndrome defined by loss of ovarian activity before the age of 40 years. The POI guideline development group of ESHRE recommends the following diagnostic criteria: oligo/ amenorrhea for at least 4 months and an elevated follicle stimulating hormone (FSH) level >25 mIU/mL on two occasion >4 weeks apart. Some clinicians and researchers proposed that POI was a progressive disease and there were three stages of POI: occult POI, biochemical POI, overt POI. However, there is lack of reliable indicators to assess the different stages of POI. The present study is to explore the change of menstruation condition, basal follicle-stimulating hormone, anti-müllerian hormone and antral follicle count during the development of POI, and whether those marks can assess the different stages of POI.

ELIGIBILITY:
Inclusion Criteria:

* Serum FSH levels ≥10mIU/ml/ serum AMH levels ≤1.0pg/ml/ AFC ≤5, on at least two occasion >4 weeks apart

Exclusion Criteria:

* Polycystic Ovarian Syndrome
* other causes of amenorrhea

Ages: 12 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients of occult premature ovarian insufficiency
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
the change of serum follicle-stimulating hormone levels | Every 3 months from date of recruit until the date of study completion, assessed up to 48 months
  the serum FSH levels between day 2 to day 5 of menstrual cycle
the change of menstruation situation | Every 3 months from date of recruit until the date of study completion, assessed up to 48 months
  Menstrual cycle
the change of serum anti-mullerian hormone levels | Every 3 months from date of recruit until the date of study completion, assessed up to 48 months
  the serum anti-mullerian hormone levels between day 2 to day 5 of menstrual cycle
the change of antral follicle count | Every 3 months from date of recruit until the date of study completion, assessed up to 48 months
  Antral follicle count between day 2 to day 5 of menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Shiling Chen, M.D./Ph.D., Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Center for Reproductive Medicine, Department of Gynecology and Obstetrics, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Society for Human Reproduction and Embryology (ESHRE) Guideline Group on POI; Webber L, Davies M, Anderson R, Bartlett J, Braat D, Cartwright B, Cifkova R, de Muinck Keizer-Schrama S, Hogervorst E, Janse F, Liao L, Vlaisavljevic V, Zillikens C, Vermeulen N. ESHRE Guideline: management of women with premature ovarian insufficiency. Hum Reprod. 2016 May;31(5):926-37. doi: 10.1093/humrep/dew027. Epub 2016 Mar 22. PMID 27008889
- [Background] Welt CK. Primary ovarian insufficiency: a more accurate term for premature ovarian failure. Clin Endocrinol (Oxf). 2008 Apr;68(4):499-509. doi: 10.1111/j.1365-2265.2007.03073.x. Epub 2007 Oct 29. PMID 17970776